CLINICAL TRIAL: NCT00021372
Title: Phase II Study of Paclitaxel and Estramustine Phosphate in Patients With Relapsed Non-Hodgkin's Lymphoma
Brief Title: Paclitaxel and Estramustine in Treating Patients With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068773; P30CA006927 (NIH); FCCC-96026; NCI-G01-1986
Record Dates: First submitted 2001-07-11; First posted 2004-02-27 (Estimated); Last update posted 2013-07-10 (Estimated); Status verified 2013-07

CONDITIONS: Lymphoma
Keywords: recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; recurrent mantle cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Estramustine; Paclitaxel

INTERVENTIONS:
Drug: estramustine phosphate sodium
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining more than one drug may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combining paclitaxel and estramustine in treating patients who have relapsed or refractory non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the response rate, time to treatment failure, and overall survival of patients with relapsed or refractory non-Hodgkin's lymphoma treated with paclitaxel and estramustine. II. Determine the toxicity of this regimen in this patient population.

OUTLINE: Patients receive oral estramustine 2-3 times daily on days 1-3 and paclitaxel IV over 1 hour on day 2 on weeks 1-6. Treatment repeats every 8 weeks for at least 1 course in the absence of disease progression or unacceptable toxicity. Patients achieving a complete or partial response continue therapy for at least 3 courses or for 1 course after achieving maximum response. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 18-35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed relapsed or refractory intermediate, high-grade, or transformed non-Hodgkin's lymphoma Received 1-3 prior treatment regimens (cytoreductive chemotherapy followed by high-dose therapy with stem cell support considered 1 regimen) Measurable disease A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Granulocyte count greater than 1,500/mm3* Platelet count greater than 75,000/mm3* * Unless due to lymphomatous marrow involvement Hepatic: Bilirubin less than 1.5 mg/dL* SGOT/SGPT less than 2 times normal* * Unless due to lymphomatous involvement Renal: Creatinine less than 2.0 mg/dL* OR Creatinine clearance greater than 50 mL/min* * Unless due to lymphomatous involvement Cardiovascular: No active uncontrolled angina pectoris No New York Heart Association class II-IV heart disease No myocardial infarction within the past 6 months No history of recurrent deep venous thrombosis not associated with catheter placement Other: No other prior malignancy within the past 5 years except curatively treated cervical cancer or basal cell or squamous cell skin cancer No serious concurrent medical illness that would preclude study No active infection

PRIOR CONCURRENT THERAPY: Biologic therapy: See Disease Characteristics Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy and recovered No prior paclitaxel, docetaxel, or estramustine Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy and recovered Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 1996-02; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell R. Smith, MD, PhD, Study Chair — Fox Chase Cancer Center
Locations (17):
- United States (17):
  - Hunterdon Regional Cancer Center, Flemington, New Jersey
  - Kimball Medical Center, Lakewood, New Jersey
  - South Jersey Regional Cancer Center, Millville, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital Burlington County, Mount Holly, New Jersey
  - Riverview Medical Center - Booker Cancer Center, Red Bank, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - St. Francis Medical Center, Trenton, New Jersey
  - Bon Secours-Holy Family Health System, Altoona, Pennsylvania
  - Delaware County Memorial Hospital, Drexel Hill, Pennsylvania
  - Pinnacle Health Hospitals, Harrisburg, Pennsylvania
  - Conemaugh Memorial Hospital, Johnstown, Pennsylvania
  - Saint Mary Regional Center, Langhorne, Pennsylvania
  - North Penn Hospital, Lansdale, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Pottstown Memorial Regional Cancer Center, Pottstown, Pennsylvania
  - Reading Hospital and Medical Center, Reading, Pennsylvania